CLINICAL TRIAL: NCT06680297
Title: A Pilot Study on Preoperative Carbohydrate Loading in Adolescent Idiopathic Scoliosis Surgery: the Impact on Safety and Enhanced Recovery
Brief Title: Preoperative Carbohydrate Drink in Adolescent Idiopathic Scoliosis Surgery: the Impact on Safety and Enhanced Recovery
Acronym: CARBO-AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1234
Record Dates: First submitted 2024-10-11; First posted 2024-11-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrates loading (Active Comparator): Participants will be given 10mls/kg of Nestle Resource carbohydrates drink a night before operation and 5mls/kg of Nestle Resource carbohydrates drink 2 hrs before operation
  Interventions: Dietary Supplement: Carbohydrates loading
- Control group (Placebo Comparator): Participants will undergo standard 6 hrs fasting with 2hr clear water before operation
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Carbohydrates loading — Patient who is randomised in the intervention group will receive Nestle drink 2hours before the operation and a night before operation. They will receive 10mls/kg a night before operation and 5mls/kg 2 hour before operation of the carbohydrate drink.
  Arms: Carbohydrates loading
Dietary Supplement: Control group — Patient assigned to this group will receive standard surgical fasting treatment which include 6hrs of fasting and 2 hrs of clear fluid prior operation
  Arms: Control group

SUMMARY:
The goal of this interventional study is to learn if carbohydrates loading improves overall outcome in adolescent patient undergoing scoliosis curgery

The main questions of the study are as follows:

1. Does carbohydrates loading improves gastrointestinal related problems such as improvement in return of bowel function measured by first passage of flatus, reduce constipation by patient's time to first bowel opening and reduce incidence of post post operative nausea and vommiting
2. Does carbohydrates loading reduces length of hospital stay and patient's overall condition in term of anxiety, thirst and hunger
3. Does carbohydrates loading affects gastric residual volume by measuring residual gastric volume with ultrasound

DETAILED DESCRIPTION:
Preoperative carbohydrate loading is strongly recommended by ESPEN as part of the clinical nutrition in surgery guideline. However, the implementation in clinical setup halted due to several limitations such as cost consuming, unfamiliar with new protocol and lack of expertise. Furthermore, there are no studies for preop carbohydrate loading in AIS as most preop carbohydrate loading is administered as a package for ERAS protocol. Thus, a strong level of evidence is necessary to propel a change in practice. As such, it is important to establish the relationship between carbohydrate loading before surgery and the impact on perioperative outcome.

Understanding the potential benefits of this nutritional intervention in the adolescent scoliosis population could contribute to the ongoing efforts to optimize surgical care in these patients. Although preoperative carbohydrates loading has strong recommendation in spinal fusion ERAS protocol, the level of evident is still scarce, more so in idiopathic scoliosis. In a systematic review, it has also stated that its limitation as most of the literature is largely retrospective studies with non-randomised data and cohort studies lacking formal control groups (Gadiya et al., 2021). Moreover, evidence on other benefits for carbohydrates loading in scoliosis surgery is still lacking such as its impact on pain, return of bowel function and post op nausea and vomiting.

This prospective study seeks to fill this knowledge gap by evaluating the influence of preoperative carbohydrate loading on postoperative outcomes in adolescents undergoing scoliosis surgery. We hypothesize that preoperative carbohydrate loading will be associated with an expedited return of bowel function, a reduced incidence of PONV, a shorter length of hospital stays, improvement in patient general wellbeing and no risk for aspiration. The objectives of this study are threefold. The primary goal of our study is to identify whether there is a significant improvement in the return of bowel function measured by flatus, reducing constipation by days of bowel opening and incidence of postoperative nausea and vomiting for patients receiving carbohydrate loading in comparison with patient that do not receive carbohydrate loading. Secondary objective also include carbohydrate loading and its effect on reducing length of hospital stay undergoing scoliosis surgery as well as patient overall condition in term of thirst, hunger and lethargy. The third objective is to measure the residual gastric volume using ultrasound before induction of anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with idiopathic scoliosis undergoing single-staged posterior spinal fusion
* Age between 10 to 19 years old
* ASA 1 & 2

Exclusion Criteria:

* Patient diagnosed with diabetes mellitus (either type I or type II)
* Patient with intellectual disability
* American Society of Anesthesiologists (ASA) class 3 and above
* Significant risk of aspiration (diagnosed with hiatal hernia, presence of GERD, BMI > 35 kg/m2 , poor GCS, swallowing abnormality, gastrointestinal abnormality)

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in bowel function by measuring days of first flatus | From post operation till patient discharge from hospital up to 1 week
  Numbers of days when patient has start passing flatus post operation
Improvement in constipation | From post operation till patient discharge from hospital up to 1 week
  The number of day when patient start to pass motion after operation
Post op nausea vomiting | Post operation within 48hours
  number of nausea and vomiting

SECONDARY OUTCOMES:
Length of hospital stay | From post operation till patient discharge from hospital up to 1 week
  How many days patient stay in hospital after operation
anxiety, thirst, hunger | Before induction of anaesthesia
  VAS score in operation theatre

OTHER OUTCOMES:
Gastric residual volume | Before induction of anaesthesia
  Ultrasound measurement of gastric residual volume pre- induction

CONTACTS AND LOCATIONS:
Overall Officials: Siti Nadzrah B Yunus, MBBS, Principal Investigator — Universiti Malaya
Locations (2):
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya, Pantai Valley, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No